CLINICAL TRIAL: NCT03459846
Title: A Phase II, Randomized, Multi-Center, Double-Blind, Comparative Global Study to Determine the Efficacy and Safety of Durvalumab in Combination With Olaparib for First-Line Treatment in Platinum-Ineligible Patients With Unresectable Stage IV Urothelial Cancer
Brief Title: A Study of Durvalumab Alone and Durvalumab+Olaparib in Advanced, Platinum-Ineligible Bladder Cancer (BAYOU)
Acronym: BAYOU
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D933IC00003; 2017-004556-27 (EudraCT Number)
Record Dates: First submitted 2018-02-22; First posted 2018-03-09 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Durvalumab/Placebo (Experimental): Durvalumab 1500 mg intravenous (IV) every 4 weeks (q4w) starting on week 1 day 1/Placebo orally (PO) twice a day (BID) starting on week 1 day 1.
  Interventions: Drug: Durvalumab; Drug: Placebo
- Arm 2: Durvalumab/Olaparib (Experimental): Durvalumab 1500 mg IV q4w starting on week 1 day 1/Olaparib PO 300 mg BID adjusted based on patient's creatinine clearance.
  Interventions: Drug: Durvalumab; Drug: Olaparib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg IV q4w
Drug: Olaparib — Olaparib PO 300 mg BID adjusted based on patient's creatinine clearance.
  Arms: Arm 2: Durvalumab/Olaparib
Drug: Placebo — Matching placebo for oral tablet BID
  Arms: Arm 1: Durvalumab/Placebo

SUMMARY:
A Phase II, Randomized, Multi-Center, Double-Blind, Comparative Global Study to Determine the Efficacy and Safety of Durvalumab in Combination With Olaparib for First-Line Treatment in Platinum-Ineligible Patients With Unresectable Stage IV Urothelial Cancer

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo controlled, multi-center, comparative global study to determine the efficacy and safety of durvalumab + olaparib combination therapy versus durvalumab + placebo (durvalumab monotherapy) as first-line treatment in patients ineligible for platinum-based chemotherapy with unresectable Stage IV urothelial cancer (UC).

ELIGIBILITY:
Inclusion criteria:

1. Provision of signed and dated, written ICF
2. Histologically or cytologically documented TCC/UC of the urothelium (including renal pelvis, ureters, urinary bladder, and urethra) also meeting the following: Unresectable, Stage IV disease; No prior systemic therapy for unresectable, Stage IV disease.
3. Ineligible for platinum-based chemotherapy defined as (i) in the opinion of the Investigator, unfit for carboplatin-based chemotherapy and (ii) meeting one of the following criteria: CrCl <60 mL/min calculated by Cockcroft-Gault equation; Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 audiometric hearing loss (25 dB in 2 consecutive wave ranges); CTCAE Grade ≥2 peripheral neuropathy; New York Heart Association Class III heart failure; ECOG 2.
4. Known tumor HRR mutation status prior to randomization.
5. World Health Organization (WHO)/ECOG performance status of 0, 1, or 2.
6. Patients with at least 1 RECIST 1.1 target lesion at baseline.
7. Ability to swallow oral medications.
8. Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients.

Exclusion criteria

1. Active or prior documented autoimmune or inflammatory disorders.
2. Other invasive malignancy within 5 years before the first dose of the IP.
3. Major surgical procedure within 28 days prior to the first dose
4. Brain metastases or spinal cord compression unless the patient's condition is stable and off steroid for at least 14 days
5. History of active primary immunodeficiency.
6. Active infection including tuberculosis (TB)
7. History of allogenic organ transplantation.
8. Uncontrolled intercurrent illness
9. Prior exposure to a PARP inhibitor or immune-mediated therapy.
10. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.
11. Current or prior use of immunosuppressive medication within 14 days before the first dose of the IP.
12. No radiation therapy is allowed, unless it is (1) definitive radiation that had been administered at least 12 months prior; (2) palliative radiation to the brain, with associated criteria for stability or lack of symptoms; or (3) palliative radiation to painful bony lesions (this must comprise less than 30% of the bone marrow) or symptomatic pelvic soft tissue mass(es).
13. Receipt of live attenuated vaccine within 30 days prior to the first dose of the IP.
14. Patients with a known hypersensitivity to durvalumab, olaparib, or any of the excipients of the products.
15. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab and 6 months for participants taking also Olaparib in case of female participants, 90 days after receipt of the last dose of the IP in case of male participants.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rosenberg, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Mark Lanasa, MD, Study Director — One MedImmune Way,Gaithersburg,Maryland,United States
Locations (34):
- United States (12):
  - Research Site, Birmingham, Alabama
  - Research Site, Goodyear, Arizona
  - Research Site, Fort Myers, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Tacoma, Washington
- Canada (5):
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Russia (4):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Rosenberg JE, Park SH, Kozlov V, Dao TV, Castellano D, Li JR, Mukherjee SD, Howells K, Dry H, Lanasa MC, Stewart R, Bajorin DF. Durvalumab Plus Olaparib in Previously Untreated, Platinum-Ineligible Patients With Metastatic Urothelial Carcinoma: A Multicenter, Randomized, Phase II Trial (BAYOU). J Clin Oncol. 2023 Jan 1;41(1):43-53. doi: 10.1200/JCO.22.00205. Epub 2022 Jun 23. PMID 35737919
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933IC00003&attachmentIdentifier=8d6faf92-3c8b-4df1-aff9-daa0d4bdddca&fileName=D933IC00003_CSP-v4_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933IC00003&attachmentIdentifier=7c54d3e7-0ea2-413a-b627-e286647898cd&fileName=D933IC00003_SAP-ed-3_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933IC00003&attachmentIdentifier=0f78e3a0-0b0b-4785-8f8b-3a6cad97c3e1&fileName=D933IC00003_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Durva + Olaparib: Patients received a combination of durvalumab 1500mg intravenous (IV) every 4 weeks (q4w) with olaparib 300mg orally (PO) twice daily (BID) adjusted based on patient's creatinine clearance
- Durva + Placebo: Patients received durvalumab 1500mg IV q4w and placebo PO BID
Period: Overall Study
Arm/Group | Durva + Olaparib | Durva + Placebo
Started | 78 | 76
Completed | 0 | 0
Not Completed | 78 | 76
Not completed — Death | 52 | 46
Not completed — Study terminated by sponsor | 24 | 28
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durva + Olaparib | Durva + Placebo | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.4 (10.8) | 70.2 (10.26) | 71.9 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 56 | 55 | 111
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 75 | 73 | 148

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival based on investigator assessments according to RECIST 1.1
Time Frame: Assessments performed at baseline and every 8 weeks from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), assessed up to the data cut-off date (15 Oct 2020), up to a max. of 31 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durva + Olaparib | Durva + Placebo
Number analyzed (Participants) | 78 | 76
Months | 4.2 [3.6 to 5.6] | 3.5 [1.9 to 5.1]
Statistical Analysis 1: Comparison: Durva + Olaparib vs Durva + Placebo; Test type: Superiority; p = 0.789, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.641 to 1.387]

2. Secondary Outcome: Overall Survival (OS)
Description: Number of Participants with Overall Survival (OS), where OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: From the date of randomization until the death due to any cause, assessed up to the data cut-off date (15 October 2020), to a maximum of 31 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Durva + Olaparib | Durva + Placebo
Number analyzed (Participants) | 78 | 76
Participants
  Died | 52 | 46
  Censored (includes subjects with unknown survival status or subjects who were lost to follow up) | 26 | 30
Statistical Analysis 1: Comparison: Durva + Olaparib vs Durva + Placebo; Test type: Superiority; p = 0.728, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.719 to 1.606]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR (per RECIST 1.1 using Investigator assessments) is defined as the number (%) of patients with at least 1 visit response of complete response (CR) or partial response (PR). CR was defined as the disappearance of all target and non-target lesions; PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters
Time Frame: From the date of randomization to the date of progression or the last evaluable assessment in the absence of progression, assessed up to the data cut-off date (15 October 2020), to a maximum of 31 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Durva + Olaparib | Durva + Placebo
Number analyzed (Participants) | 78 | 76
Participants
  Response | 22 | 14
  No Response | 56 | 62
Statistical Analysis 1: Comparison: Durva + Olaparib vs Durva + Placebo; Test type: Superiority; p = 0.142, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.821 to 3.778]

4. Secondary Outcome: Duration of Response (DoR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DoR is the time from the date of first documented response until the date of documented progression or death in the absence of disease progression
Time Frame: Tumor assessments every 8 weeks after randomization for the first 48 weeks and then every 12 weeks thereafter until the date of objective disease progression. Assessed up to the data cut-off date (15 October 2020), to a maximum of 31 months
Population: Duration of Response (DoR) was calculated for all responders (N=36)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Durva + Olaparib | Durva + Placebo
Number analyzed (Participants) | 22 | 14
Months | 8.9 [4.7 to 12.1] | 14.8 [7.5 to 17.2]

ADVERSE EVENTS:
Time Frame: From first administration of study treatment until 90 days after the last dose of study medication, assessed up to the data cut-off date (15 October 2020), to a maximum of 31 months
Description: There were 78 subjects randomised to Durva + Olaparib (Full Analysis Set), however 2 of these subjects did not receive treatment (resulting in 76 in the Safety Analysis Set). Hence, for Durva + Olaparib, the Total number at risk for all-cause mortality = 78 while the Total # at Risk by any Serious Adverse Event = 76 and the Total # at Risk by any Other Adverse Event = 76
Arm/Group | Durva + Olaparib | Durva + Placebo
All-Cause Mortality (participants affected / at risk) | 52/78 | 46/76
Serious Adverse Events (participants affected / at risk) | 37/76 | 26/76
Other Adverse Events (participants affected / at risk) | 65/76 | 63/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva + Olaparib (N=76) | Durva + Placebo (N=76)
Urinary tract infection (Infections and infestations) | 6 (7) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (5) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva + Olaparib (N=76) | Durva + Placebo (N=76)
Anaemia (Blood and lymphatic system disorders) | 34 (50) | 21 (22)
Hypothyroidism (Endocrine disorders) | 7 (7) | 4 (5)
Nausea (Gastrointestinal disorders) | 20 (23) | 6 (6)
Constipation (Gastrointestinal disorders) | 13 (14) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 5 (7)
Vomiting (Gastrointestinal disorders) | 7 (8) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 22 (25) | 13 (13)
Asthenia (General disorders) | 10 (11) | 2 (2)
Pyrexia (General disorders) | 7 (7) | 7 (9)
Oedema peripheral (General disorders) | 3 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 9 (11) | 4 (4)
Blood creatinine increased (Investigations) | 8 (9) | 4 (4)
Amylase increased (Investigations) | 4 (5) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 19 (22) | 10 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 4 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 7 (8) | 6 (6)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8)
Hypertension (Vascular disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03459846/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03459846/SAP_001.pdf